CLINICAL TRIAL: NCT05376514
Title: Investigation Into the Effects of Central Blood Pressure Variability and Antihypertensive Adherence on the Size and Growth Rate of Abdominal Aortic Aneurysms
Brief Title: Central Blood Pressure and Variability Evaluation
Acronym: CAVE-ON
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22SM7440
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: AAA; Abdominal Aortic Aneurysm; Blood Pressure
Keywords: AAA; Central blood pressure; Growth; Medication adherence; Blood pressure variability
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: A sub-study of the AARDVARK (Aortic Aneurysmal Regression of Dilation: Value of ACE-Inhibition on RisK) trial indicated a statistically significant association between central blood pressure (BP) variability and abdominal aortic aneurysm (AAA) growth. The role of anti-hypertensive adherence has not been explored in the context of AAA growth.

Objective: To confirm whether higher central BP variability is associated with higher AAA growth rates and to examine the effect of medication adherence on AAA growth rates in a prospective longitudinal cohort study.

Methods: Up to 175 patients will be recruited over ten months from two sites with standardised quality control of AAA, BP and antihypertensive non-adherence measurement. Patients (>55 years), with AAAs ≥3cm in diameter (including AAA ≥5.5cm, not proceeding to surgery) will be recruited and undergo AAA ultrasound (US), BP (peripheral and central) and antihypertensive non-adherence measurements every four months (+/- one month) for 24 months. Ambulatory BP variability data will be collected. Data on medication adherence and beliefs around medications will be collected with validated questionnaires.

Analysis: Primarily, the relationship between central diastolic BP visit-to-visit variability and AAA growth (estimated by multilevel modelling) based on US measurements and secondarily the relationship between central diastolic BP variability and time taken to reach the threshold for AAA repair (5.5 cm) or rupture.

DETAILED DESCRIPTION:
The AARDVARK (Aortic Aneurysmal Regression of Dilation: Value of ACE-Inhibition on RisK) trial was designed to investigate the hypothesis that an ACE-inhibitor (perindopril) would reduce growth rate of small AAAs in a three-arm randomised placebo-controlled trial. While this didn't show a significant effect, results from an in-trial sub-study (CAVE study) demonstrated a significant relationship between central BP variability and aneurysm growth rates. This requires confirmation, in a dedicated study.

Design:

This is a multicentre prospective longitudinal observational cohort study. Each patient will have a study visit every 4 months with a minimum of 6 clinical visits where the study team will collect demographic data; psychological data (short form questionnaires that can be independently filled in); and physical data. The study team will also access routinely collected NHS cross-sectional imaging for comparison throughout the study, as quality control. No additional procedures involving ionising radiation will take place.

Study timeline:

There will be a 10-month recruitment period; all subjects will attend visits for a period of 18-24 months. The data collection will continue for 24 months in total. There will be a 6-month period of data analysis and write up.

Recruitment:

A cohort of up to 175 patients will be recruited from two trusts in London comprising four hospitals - Imperial College Healthcare NHS Trust (ICH) at St Mary's and Charing Cross hospitals, and London North West University Healthcare Trust (LNWH) at Northwick Park and Hillingdon hospitals. All visits and measurements will take place at central sites (St Mary's and Northwick Park hospitals).

Data Collection:

1. Demographic data - e.g. current prescribed anti-hypertensive medication and other cardiovascular medications, height and weight, medical history, smoking status
2. Psychological data - three short-form questionnaires that can be independently filled in by participants. Questionnaires will constitute measures of anxiety and depression (Hospital Anxiety and Depression Score [HADS]), current medication adherence (modified Voils Adherence Score), and beliefs around medication and adherence (Beliefs about Medicines Questionnaire [BMQ]).
3. Physical data - sitting mean peripheral and central systolic and diastolic BP, visit-to-visit central systolic and diastolic BP variability measured as standard deviation, coefficient of variation and variation independent of the mean will be measured using a validated arm cuff-based method. Ambulatory BP parameters will be measured using a validated monitor. USS AAA measurement will take place at bedside in supine position with outer-to-outer (OTO) calliper placement.

Primary Endpoint Analysis:

The association between central BP variability measured as standard deviation and AAA growth will be analysed using regression models where BP variability is the exposure and AAA growth is the outcome.

Random effects multilevel models where level-1 units are AAA repeated measurements nested within patients (level-2 units) will be used to estimate AAA growth. To explore non-linearity in AAA growth appropriate modelling will be used eg. linear splines.

Secondary Endpoints Analyses:

Survival analysis techniques such as Cox proportional hazards models will be used to assess the relationship between central BP variability and time taken for the AAA to reach the threshold for intervention (5.5 cm) or rupture.

Associations between haemodynamic parameters and aneurysm growth rate will be investigated. For each of the other measurements of systolic and diastolic central BP variability (coefficient of variation (SD ÷ mean) and variation independent of the mean calculated as SD÷(mean x) where x is determined empirically by curve fitting) and for other BP and haemodynamic parameters studied, the same multilevel model or generalised linear models will be used to estimate AAA growth. All analyses will be adjusted for an a-priori list of confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* infrarenal aneurysms of ≥3cm in size (to include AAA ≥5.5cm in those not proceeding to surgery)

Exclusion Criteria:

* Patient's with a known genetic aetiology of their AAA
* age<55
* known bilateral proximal upper extremity obstructive lesions
* persistent cardiac arrhythmia
* those unable to give informed consent
* those too frail to travel for four monthly surveillance
* any clinically significant medical condition which, in the opinion of the investigator, may interfere with the study results and/or reduce life expectancy to < 2 years
* participation in another trial of an investigational product or device within the previous 30 days
* unable or unwilling to comply with the requirements of the study, in the opinion of the investigator

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an AAA currently under surveillance, or those with an AAA ≥5.5cm not proceeding to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Growth | 24 months
  AAA growth as measured by multilevel modelling

SECONDARY OUTCOMES:
Time to rupture or repair | 24 months
  Time taken for patient's AAA to rupture or to reach threshold for repair

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Northwick Park Hospital, London North West Healthcare NHS Trust, London
  - St Mary's Hospital, Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Undecided